CLINICAL TRIAL: NCT03802656
Title: Safety and Feasibility of a Vertebral Body Tethering Technique for Pediatric Idiopathic Scoliosis
Brief Title: Vertebral Body Tethering Treatment for Idiopathic Scoliosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device is no longer investigational. It has been approved by the FDA as an HUD under HDE H190005.
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: VBT120718
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Scoliosis; Spinal Curvatures; Spinal Diseases; Bone Diseases; Musculoskeletal Disease; Adolescent Idiopathic Scoliosis; Juvenile; Scoliosis
Keywords: Scoliosis; Idiopathic Scoliosis; Adolescent Idiopathic Scoliosis; Vertebral Body Tethering; growth modulation spine; spine; juvenile scoliosis
MeSH Terms: conditions — Scoliosis; Spinal Curvatures; Spinal Diseases; Bone Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Anterior Vertebral Body Tethering (Experimental): Subjects who will be undergoing the anterior vertebral body tethering surgery.
  Interventions: Device: Anterior Vertebral Body Tethering

INTERVENTIONS:
Device: Anterior Vertebral Body Tethering — Vertebral body tethering through anterior thoracoscopic approach under general anesthesia and fluoroscopic guidance.

SUMMARY:
This study will determine whether vertebral body tethering is a safe and feasible method of treatment for pediatric idiopathic scoliosis.

DETAILED DESCRIPTION:
Scoliosis is a condition in which the spine is deformed by a curvature in the coronal plane. It is generally associated with a twisting (axial plane) deformity as well. It can have a variety of underlying etiologies and the etiology is used to classify the types of scoliosis. Idiopathic scoliosis is sub-classified in two ways: by age of onset and by magnitude of deformity. Curves between 10 and 25 degrees are considered mild. Curves between 25 and 50 degrees are classified as moderate. Curves greater than 50 degrees are termed severe. The current standard of care for moderate scoliosis in patients with remaining growth is to utilize a thoracolumbosacral orthosis (TLSO brace) to prevent progression of deformity. The scientific evidence has supported the efficacy of this intervention in avoiding progression of the Cobb angle to 50 degrees or more.

If treated with a TLSO brace, many idiopathic scoliosis patients would conceivably be subjected to years of brace wear and the cost and psychological factors inherent therein. Additional downsides of brace treatment include the potentially negative psychosocial impact of wearing an external sign of deformity during adolescence, a key period of emotional development. Prior research has identified negative psychosocial effects related to wearing a brace in children.

Recent evidence has suggested that certain curve patterns will likely progress to 50 degrees or more, despite treatment with a TLSO brace. Sanders, et al. demonstrated a correlation of Cobb angle (greater than 35 degrees) and skeletal maturity (bone age 4 or less) to the risk of progression to 50 degrees or more, despite TLSO bracing. The evidence supports that the current practice of TLSO bracing is not an effective treatment to avoid progression to 50 degrees in these patients. It is on this population (thoracic Cobb angle greater than 35 degrees, bone age of 4 or less) that we intend to test the safety and feasibility of Anterior Vertebral Body Tethering to avoid curve progression to 50 degrees.

The study intervention is surgical orthopedic implantation of the Anterior Vertebral Tether Device, by way of thoracoscopic surgery under general anesthesia. The primary outcome measures include assessments of safety of the insertion procedure and of the device, as well as the secondary measure of feasibility by determining the ability to successfully implant the investigational device.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 8 to 16 years old at time of enrollment (inclusive)
2. Diagnosis of idiopathic scoliosis
3. Sanders bone age of less than or equal to 4
4. Thoracic or thoracolumbar/lumbar curves of greater than or equal to 35 degrees and less than or equal to 60 degrees from levels T4 through L3
5. Lenke classification of 1, 2, 3, 5, or 6
6. Patient has already been identified for and recommended to have surgical intervention
7. Spina bifida occulta is permitted
8. Spondylolysis or Spondylolisthesis is permitted, as long as it is non-operative, the patient has not had any previous surgery for this, and no surgery is planned in the future
9. Completed standard-of-care procedures as outlined in Section 5

Exclusion Criteria:

1. Pregnancy (current)
2. Prior spinal or chest surgery
3. MRI abnormalities (including syrinx greater than 4mm, Chiari malformation, or tethered cord)
4. Neuromuscular, thoracogenic, cardiogenic scoliosis, or any other non-idiopathic scoliosis
5. Associated syndrome, including Marfan Disease or Neurofibromatosis
6. Sanders bone age greater than 4
7. Thoracic or thoracolumbar/lumbar curves less than 35 degrees or greater than 60 degrees
8. Compensatory curve greater than 35 degrees without intent to treat surgically
9. Unable or unwilling to firmly commit to returning for required follow-up visits
10. Investigator judgement that the subject/family may not be a candidate for the intervention

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of Treatment-Emergent Adverse Events | 2 years after last subject's device implantation
  Intraoperative and post-intervention medical events or signs and symptoms of complications arising after the start of study intervention will be captured. The event description, date of onset, end date, severity, and outcome will be documented. The frequencies, type, body system, severity, and relationship to the study intervention will also be summarized. A distinction will be made between those events which are "device-related" and "non device-related".

SECONDARY OUTCOMES:
Feasibility: Incidence of Successfully Implanted Tether Devices | 2 years after last subject's device implantation
  The feasibility of the vertebral body tethering device will analyzed based on successful implantation of the device. Implantation will be considered a failure if the device breaks/loosens after implantation, or if it overcorrects the spinal curve.
Efficacy: Comparison of Preoperative and Postoperative Cobb Angle | 2 years after last subject's device implantation
  The exploratory therapeutic endpoint used for feasibility will be change in post-operative Cobb angle compared to pre-operative Cobb angle, measured on coronal radiograph of the spine.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Haber, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Health System- Jefferson Hwy, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No